CLINICAL TRIAL: NCT05620381
Title: Health and Sleep Assessment After the Strasbourg Attacks of December 11, 2018
Acronym: ELSSAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7713
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-11

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders; Disorders Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the prevalence of post-traumatic stress disorder (PTSD), associated risk factors, health care consumption, and sleep disorders in a civilian population exposed to the December 11, 2018, attacks in Strasbourg. Terrorist attacks have unfortunately become all too frequent on our territory in recent years. A better knowledge of the psychological and psychiatric repercussions on exposed populations is essential in order to better prevent and treat disorders that can have a major functional impact on the lives of exposed individuals and to adapt care during future similar events

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥ 18 years old),
* Having been exposed to the attacks of December 11, 2018 in Strasbourg directly or indirectly (presence at the scene or close relative present at the scene)
* Subject who has not expressed his opposition, after information, to the reuse of his data for the purpose of this research

Exclusion Criteria:

* Subject who has expressed opposition to participating in the study
* Subject under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) having been exposed to the attacks of December 11, 2018 in Strasbourg directly or indirectly (presence at the scene or close relative present at the scene)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective evaluation of the prevalence of post-traumatic stress disorder (PTSD) in a population exposed to the attacks of December 11, 2018 in Strasbourg | Files analysed retrospectively from February 11, 2018 to November 30, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie d'Urgences, de Liaison et de Psychotraumatologie - CHU de Strasbourg - France, Strasbourg, France